CLINICAL TRIAL: NCT05884229
Title: The Effect of SPI (Surgical Pleth Index) - Guided Anaesthesia Versus Conventional Analgesia on Opioid Consumption Under Multimodal Analgesia in Gastric Sleeve Surgery
Brief Title: The Effect of SPI (Surgical Pleth Index) - Guided Anaesthesia on Opioid Consumption in Gastric Sleeve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Leahu Crina, MD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Intraoperative Monitoring
Keywords: nociception monitoring; SPI; opioid consumption; gastric sleeve; analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard opioid administration (No Intervention)
- SPI-guided opioid administration (Experimental)
  Interventions: Other: Intra-operative analgesia guided by SPI

INTERVENTIONS:
Other: Intra-operative analgesia guided by SPI — In the SPI-guided group, when SPI is higher than 50 for the first time and for more than 3 minutes, we will administer 1,0 μg/kg of fentanyl LBW. When SPI is again higher than 50 and for more than 5 minutes, we will re-administer 1,0 μg/kg of fentanyl LBW. We will repeat until SPI is between 20-50.
  Arms: SPI-guided opioid administration

SUMMARY:
This is a unicentric, prospective randomised trial that aims to evaluate the role of intra-operative monitoring of nociception through SPI (Surgical Pleth Index) in guiding analgesia and reducing opioid consumption in obese patients undergoing bariatric surgery.

We aim to enrol 40 patients having laparoscopic gastric sleeve surgery in the Cluj-Napoca County Hospital. They will be randomised into two groups, one with opioid administration during surgery guided by SPI, and the other one guided by anesthetist experience. We will monitor opioid consumption, pain scores during the first 90 minutes post-operatively, hemodinamic events during surgery and the duration between reversal of neuromuscular block and extubation.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to laparoscopic gastric sleeve surgery in First Surgical Clinic, Cluj-Napoca County Hospital

Exclusion Criteria:

* drugs that affect the autonomic nervous system
* peripheral neuropathy
* altered renal/hepatic function
* chronic opioid use
* use of vaso-active drugs intra-operatively

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores on the visual analog scale during the first 90 minutes post-operatively | during the first 90 minutes post-operatively
  Pain scores on the visual analog scale during the first 90 minutes post-operatively

SECONDARY OUTCOMES:
Opioid consumption | during surgery
  the amount of fentanyl per LBW
Sevoflurane concentration | during surgery
  mean MAC and sevoflurane concentration during surgery
Time from neuromuscular reversal to extubation | at the end of surgery
  Time from neuromuscular reversal to extubation
Hemodinamic events | during surgery
  an increase in heart rate or mean arterial pressure with more than 20% of the basal values (measured on the ward)
Rescue analgesia | in the first 90 minutes post-operatively
  the need for rescue opioids during the first 90 minutes post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- First Surgical Clinic, County Hospital, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ledowski T, Schneider M, Gruenewald M, Goyal RK, Teo SR, Hruby J. Surgical pleth index: prospective validation of the score to predict moderate-to-severe postoperative pain. Br J Anaesth. 2019 Aug;123(2):e328-e332. doi: 10.1016/j.bja.2018.10.066. Epub 2019 Mar 12. PMID 30916030
- [Background] Chen X, Thee C, Gruenewald M, Ilies C, Hocker J, Hanss R, Steinfath M, Bein B. Correlation of surgical pleth index with stress hormones during propofol-remifentanil anaesthesia. ScientificWorldJournal. 2012;2012:879158. doi: 10.1100/2012/879158. Epub 2012 Sep 2. PMID 22973178
- [Background] Bapteste L, Szostek AS, Chassard D, Desgranges FP, Bouvet L. Can intraoperative Surgical Pleth Index values be predictive of acute postoperative pain? Anaesth Crit Care Pain Med. 2019 Aug;38(4):391-392. doi: 10.1016/j.accpm.2018.05.004. Epub 2018 May 29. No abstract available. PMID 29857187
- [Background] Bergmann I, Gohner A, Crozier TA, Hesjedal B, Wiese CH, Popov AF, Bauer M, Hinz JM. Surgical pleth index-guided remifentanil administration reduces remifentanil and propofol consumption and shortens recovery times in outpatient anaesthesia. Br J Anaesth. 2013 Apr;110(4):622-8. doi: 10.1093/bja/aes426. Epub 2012 Dec 5. PMID 23220856
- [Background] Chen IW, Lin CM, Chang YJ, Chen JY, Wu ZF, Ho CN, Feng IJ, Sun CK, Hung KC. Association of surgical pleth index with late postoperative analgesic requirement: A retrospective study. J Clin Anesth. 2020 Mar;60:12-13. doi: 10.1016/j.jclinane.2019.08.022. Epub 2019 Aug 19. No abstract available. PMID 31437589
- [Background] Guo J, Zhu W, Shi Q, Bao F, Xu J. Effect of surgical pleth index-guided analgesia versus conventional analgesia techniques on fentanyl consumption under multimodal analgesia in laparoscopic cholecystectomy: a prospective, randomized and controlled study. BMC Anesthesiol. 2021 Jun 4;21(1):167. doi: 10.1186/s12871-021-01366-x. PMID 34088270
- [Background] Hung KC, Huang YT, Kuo JR, Hsu CW, Yew M, Chen JY, Lin MC, Chen IW, Sun CK. Elevated Surgical Pleth Index at the End of Surgery Is Associated with Postoperative Moderate-to-Severe Pain: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2022 Sep 6;12(9):2167. doi: 10.3390/diagnostics12092167. PMID 36140567
- [Background] Won YJ, Lim BG, Kim YS, Lee M, Kim H. Usefulness of surgical pleth index-guided analgesia during general anesthesia: a systematic review and meta-analysis of randomized controlled trials. J Int Med Res. 2018 Nov;46(11):4386-4398. doi: 10.1177/0300060518796749. Epub 2018 Sep 9. PMID 30198405